CLINICAL TRIAL: NCT00797810
Title: Intensification Therapy of Mature B-ALL, Burkitt and Burkitt Like and Other High Grade Non-Hodgkin's Lymphoma in Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Giovanni Martinelli, Dipartiemento di Ematoogia "seragnoli"- Policlinico Sant'Orsola di Bologna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEMOS ALL1105
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Acute Lymphoblastic Leukemia; Non-Hodgkin's Lymphoma
Keywords: Acute lymphoblastic leukemia of the mature B-cell type; High-grade non-Hodgkin's lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin | interventions — Rituximab; Cyclophosphamide; Prednisone; Dexamethasone; Vincristine; Ifosfamide; Cytarabine; Doxorubicin; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- therapy (Experimental)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab
  Other Names: Cyclophosphamide, Prednisone, Dexamethasone, Vincristine, Ifosfamide, Cytarabine, Adriamycin, G-CSF

SUMMARY:
All patients are treated according to the same therapy regimen. Therapy duration (number of cycles) and radiotherapy vary according to age group, stage and response. Chemotherapy consists of a pre-phase-treatment (for all patients) and varying A, B and C cycles. Therapy for Patients in the 18-55 Age Group

* Patients in stages III-IV and all patients with mediastinal tumors or extranodal involvement are administered 6 cycles (A1, B1, A2, B2, A3, B3).
* Chemotherapy is stopped after 4 cycles (A1, B1, A2, B2) for patients with stage I/ II if a clear CR has been achieved and there is initially no mediastinal or extranodal involvement.
* In cases of refractory or progressive disease after 4 cycles, study therapy is stopped. These patients are to be given salvage therapy with subsequent stem cell transplantation. Therapy for Patients older than 55 years
* The course corresponds to that of patients in the younger age group, but the regimen is dose reduced (A1*, B1*,A2*, B2*, A3*, B3*). Antibody therapy with anti-CD20 is to be administered on day 1 of each chemotherapy cycle (A, B). After end of chemotherapy (6 or 4 cycles) 2 more cycles of anti-CD 20 are to be administered to reach a total number of 8 resp. 6 cycles antibody therapy.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphoblastic leukemia of the mature B-cell type (L3-ALL)
* High-grade non-Hodgkin's lymphoma of the following subtypes (WHO classification)

  * Burkitt's lymphoma (including atypical Burkitt's lymphoma)
  * Precursor B-lymphoblastic lymphoma
  * Anaplastic large-cell lymphoma (Ki1+, B-, T- oder Null-cell-type)
  * Mediastinal large B-cell-lymphoma (subtype of diffuse large B-cell lymphoma)
* Age = 18 years
* Patient's Informed Consent

Exclusion Criteria:

* Serious complications caused by leukemia/ lymphoma or by a second illness: e.g.

  * Severe, unmanageable complications such as sepsis, pneumonia with oxygen deficiency,
  * Shock, hemorrhage at the time of diagnosis
  * Renal insufficiency from leukemia/lymphoma-unrelated causes
  * Severe cardiac or hepatic insufficiency
  * Severe obstructive or restrictive lung disease that would compromise patient's treatment with intensified chemotherapy
  * HIV infection
  * Secondary lymphoma following prior chemotherapy/ radiotherapy or an active second malignancy
  * Known severe allergy to foreign proteins
* Cytostatic pretreatment for B-ALL/lymphoma (exceptions: short-term administration of steroids = 7 days, single administration of vincristine or cyclophosphamide, one cycle of CHOP, a single administration in an emergency of other cytostatic agents) for another malignant disease within the last 5 years
* Pregnancy/ nursing period
* Severe psychiatric illness or other circumstances giving ground to the assumption that a patient cannot give his consent to therapy or act co-operatively
* Absence of patient's informed consent
* Participation in another clinical study that would possibly interfere with study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2006-12

PRIMARY OUTCOMES:
Test of the tolerability and efficacy of new therapy elements to improve remission
Rates, overall survival and remission duration
Administration of anti-CD20 (rituximab ®) together with combination chemotherapy
Combination therapy with high-dose methotrexate and high-dose cytarabine together with conventional cytostatic agents (cycle C)
Prophylactic administration of G-CSF after every cycle of chemotherapy
Localised irradiation after 6 cycles in mediastinal tumor cases, CNS involvement and residual tumor

SECONDARY OUTCOMES:
Test of the age-adapted therapy stratification according to biological age
(18< age <55)
Definition of prognostic factors
Setting up of a central reference pathology panel

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Martinelli, MD, Principal Investigator — Institute of Haematology "L.e A. Seragnoli" Bologne-Italy
Locations (1):
- Institute of Haematology "L. e A. Seragnoli", Bologna, Italy